CLINICAL TRIAL: NCT01582932
Title: A Multicenter, Open-label, Phase 1 Study of the Safety, Tolerability, Systemic Exposure, Pharmacodynamics, and Treatment Effect of Calcipotriene Foam, 0.005%, in Pediatric Subjects (Ages 2 to 11 Years) With Plaque Psoriasis
Brief Title: Evaluate Safety and Tolerability of Calcipotriene Foam 0.005% in Pediatric Subjects With Mild/Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STF115469
Record Dates: First submitted 2012-03-29; First posted 2012-04-23 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; pediatric; mild; moderate
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Calcipotriene 0.005% Foam (Experimental): Foam is a vitamin D3 analog (calcipotriene) foam 0.005%. It is applied twice a day for 8 weeks to psoriasis lesions (except the face).
  Interventions: Drug: Calcipotriene 0.005% Foam

INTERVENTIONS:
Drug: Calcipotriene 0.005% Foam — All treatments will be administered topically twice daily (morning and evening) for 8 weeks to areas affected with psoriasis (excluding face).
  Other Names: Sorilux

SUMMARY:
Calcipotriene is a vitamin D3 analog that has been used as topical therapy in adult subjects with plaque-type psoriasis since 1993. Calcipotriene foam, 0.005%, was approved in 2010 for the treatment of plaque psoriasis in adults aged 18 years and older. The current study is a multicenter study evaluating calcipotriene foam, 0.005% in pediatric subjects (ages 2 to 11 years, inclusive) with mild to moderate plaque psoriasis. Subjects or their primary caregivers will apply calcipotriene foam, 0.005%, as a thin layer twice a day on the body and scalp for up to 8 weeks. The safety, tolerability, pharmacodynamics, and pharmacokinetics of calcipotriene will be evaluated.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1 study in a total of 75 pediatric subjects, ages 2 to 11 years, inclusive, with mild or moderate plaque psoriasis.

The study will enroll sufficient subjects with plaque psoriasis and an ISGA score of mild to moderate (score of 2 or 3) at Baseline to ensure 50 evaluable subjects in a general use cohort.

In addition, a sufficient number of subjects with moderate plaque psoriasis will be enrolled to ensure 25 evaluable subjects in a 'maximum-use' cohort that have:

A. At least 10% total BSA with some scalp involvement (15 evaluable subjects ages 7 to 11 years) or B. At least 3% total BSA with some scalp involvement (10 evaluable subjects ages 2 to 6 years). "Napkin" psoriasis (psoriasis in the diaper area) can be included in the BSA calculation for this age group.

Subjects or their caregivers will apply a thin layer of study product twice a day to the treatment areas for 8 weeks. Any new psoriatic lesions appearing in treatment areas during the treatment period should also be treated with study product. Safety assessments (adverse event and serious adverse event query) will occur at all study visits. Treatment effect assessments, urine calcium metabolism assessments, and application site tolerability assessments will be performed for all subjects at all in-clinic visits. A blood sample will be taken from all subjects at Screening for evaluation of pharmacodynamic (PD) and 2,5-OH vitamin D levels, an additional blood draw for PD parameters will be taken at Week 2 for the maximum-use cohort only. Blood sampling for pharmacokinetic (PK) measurements will be performed in the maximum-use cohort at Screening and Week 2.

ELIGIBILITY:
A. At least 10% total BSA with some scalp involvement (15 evaluable subjects ages 7 to 11 years) or B. At least 3% total BSA with some scalp involvement (10 evaluable subjects ages 2 to 6 years). "Napkin" psoriasis (ie, psoriasis in the diaper area) can be included in the BSA calculation for this age group.

Key Inclusion Criteria:

* Male or female subjects, ages 2 to 11 years, inclusive, at the time of consent
* For the maximum-use cohort:

A. ISGA of 3 or higher at Screening (see Appendix 2). Ages 7 to 11 - at least 10% total BSA with some scalp involvement (See Appendix 1).

Ages 2 to 6 - at least 3% total BSA (napkin psoriasis included) with some scalp involvement (See Appendix 1).

-For the general use cohort, an ISGA score of 2 or 3 at Screening with no BSA minimum.

Key Exclusion Criteria:

* Any inflammatory skin disease in the treatment area that may confound the evaluation of the plaque psoriasis
* Current diagnosis of unstable forms of psoriasis in the treatment area, including guttate, erythrodermic, exfoliative, or pustular psoriasis
* Use of any topical treatments that have a known beneficial effect on psoriasis, including but not limited to corticosteroids, retinoids, vitamin D derivatives, coal tar, tazarotene, medicated shampoos, or anthralin, within 2 weeks prior to enrollment
* Use of nonbiologic systemic antipsoriatic therapy (eg, corticosteroids, psoralen, retinoids, methotrexate, cyclosporine, other immunosuppressive agents), biologic therapy (eg, adalimumab, etanercept, golimumab, infliximab, ustekinumab), or phototherapy (eg, psoralen and ultraviolet A [PUVA], ultraviolet B [UVB]) within 4 weeks prior to enrollment
* Use of or need for initiation of any nonpsoriatic therapy that might affect psoriasis (including antimalarials, β-blockers, interferon, or lithium) within 4 weeks prior to enrollment
* Use of medications that affect or change calcium and parathyroid hormone (PTH) concentrations or interfere with the measurement of calcium or PTH concentrations within 4 weeks prior to enrollment
* Known difficult venous access beyond that expected for subject age
* Average daily ingestion of more than 2000 mg of elemental calcium or more than 1000 IU of vitamin D within 2 weeks prior to enrollment
* History of hypersensitivity, known allergy, or other adverse reaction to calcipotriene or other vitamin D analogs or to any component of the study product
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders
* Use of any investigational therapy within 4 weeks prior to enrollment
* Pregnant or breast feeding female or females who do not use contraception
* Current immunosuppression
* Albumin-adjusted serum calcium at screening that is above the upper limit of normal

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment effect and change in ISGA scores of body and scalp psoriasis (Safety and Tolerability) | 56 weeks
  To evaluate the safety and tolerability of calcipotriene foam, 0.005%, in pediatric subjects (ages 2 to 11 years, inclusive) with mild to moderate plaque psoriasis. An evaluation of treatment effect will include changes in ISGA scores of body and scalp psoriasis from baseline. Safety will be assessed based on vital signs, reported adverse events (AEs), use of concomitant medications, and application site tolerability assessments.

SECONDARY OUTCOMES:
Plasma concentrations (trough) of calcipotriene | 8 weeks
  Describe the plasma concentrations (trough) of calcipotriene following administration of foam, 0.005%, in pediatric subjects (ages 2 to 11 years, inclusive) with moderate plaque psoriasis.
Pharmacodynamic effect | 2 weeks
  To evaluate the pharmacodynamic effect (ie, calcium metabolism) of calcipotriene foam 0.005%, in pediatric subjects (ages 2 to 11 years, inclusive) with mild to moderate plaque psoriasis.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mudge, Study Director — Sponsor GmbH
Locations (34):
- United States (34):
  - Investigational Site, Birmingham, Alabama
  - Investigational Site, Rogers, Arkansas
  - Investigational Site, Encino, California
  - Fountain Valley, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Investigational Site, Hollywood, Florida
  - Investigational Site, Jacksonville, Florida
  - Miami, Florida
  - Investigational Site, Miami, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, Alpharetta, Georgia
  - Atlanta, Georgia
  - Investigational Site, Marietta, Georgia
  - Investigational Site, Sandy Springs, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Plainfield, Indiana
  - Brighton, Massachusetts
  - Investigational Site, Farmington Hills, Michigan
  - Saint Joseph, Missouri
  - Investigational Site, St Louis, Missouri
  - Investigational Site, New York, New York
  - Investigational Site, Chapel Hill, North Carolina
  - Investigational Site, Winston-Salem, North Carolina
  - Investigational Site, Portland, Oregon
  - Investigational Site, Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Investigational Site, Austin, Texas
  - Investigational Site, Houston, Texas
  - San Antonio, Texas
  - Investigational Site, Salt Lake City, Utah
  - Investigational Site, Norfolk, Virginia
  - Investigational Site, Spokane, Washington
  - Investigational Site, Tacoma, Washington